CLINICAL TRIAL: NCT03615859
Title: Objective Markers and New Indicators in Adrenal Insufficiency Disease (OMNI-AID Study)
Brief Title: Objective Markers and New Indicators in AI Disease (OMNI-AID Study)
Acronym: OMNI-AID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: 18HH4425; 216757 (Other: IRAS ID); 18/LO/0069 (Other: REC reference number)
Record Dates: First submitted 2018-07-31; First posted 2018-08-06 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Adrenal Insufficiency
Keywords: Glucocorticoids; Hydrocortisone; Prednisolone
MeSH Terms: conditions — Adrenal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum, plasma, urine and peripheral blood mononuclear cells will be stored as part of this study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Healthy volunteers: Healthy volunteers whose data represents a negative control
- Prednisolone replacement group: Participants with adrenal insufficiency who are treated with replacement doses of prednisolone
- Hydrocortisone replacement group: Participants with adrenal insufficiency who are treated with replacement doses of hydrocortisone
- New adrenal insufficiency group: Participants who have recently been given a new diagnosis of adrenal insufficiency
- High dose steroids groups: Participants who are treated with high dose steroids for management of any medical condition to serve as a positive control

SUMMARY:
This pilot study is designed to compare healthy volunteers with three groups of patients with adrenal insufficiency and a final group of patients receiving high dose steroids for anti-inflammatory purposes. The study will collect data on all 5 groups with the intention of identifying any novel markers or immunological indicators which may be used clinically to gauge the adequacy of steroid replacement treatment in patients with adrenal insufficiency.

DETAILED DESCRIPTION:
Glucocorticoid replacement in adrenal insufficiency poses a significant challenge. If given too much, patients risk long term complications including diabetes, osteoporosis and cardiovascular disease. If, however they are given too little, patients can feel tired, unwell and may collapse as there is insufficient steroid hormone to cope with stress.

Currently there is no single objective marker or outcome that can be measured to ascertain whether a patient is receiving optimum glucocorticoid replacement therapy. This study will investigate a selection of markers to examine whether they can be used to as indicators to gauge the adequacy of therapy. Finding an appropriate marker could unlock better care and outcomes for our patients with adrenal insufficiency .

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 - 85 years
* Male or female
* Participants who are otherwise healthy enough to participate, as determined by pre-study medical history and physical examination

Patient groups only:

* Diagnosed with AI for over 6 months according to standard diagnostic criteria or with a medical condition requiring acute high dose steroid therapy for anti-inflammatory purposes
* If diagnosed with AI, established on stable HC replacement or prednisolone replacement, dose not altered for at least 3 months
* Established on a stable dose of Fludrocortisone, if taking, dose not altered for at least 3 months
* Participants taking other hormone replacements (e.g. levothyroxine, testosterone or growth hormone in secondary adrenal insufficiency) are accepted providing that their replacement doses have not altered for at least 3 months
* Participants who are able and willing to give written informed consent to participate in the study.

Exclusion Criteria:

* Participants with a diagnosis of Type 1 or Type 2 diabetes mellitus.
* Unable to give informed consent.
* Excessive caffeine intake above 500 mg per day.
* Taking supplements or herbal medications that the participant is unwilling or unable to stop prior to and during the study period e.g. St John's Wort (may decrease prednisolone levels), Cat's claw, Echinacea (immunomodulatory properties).
* Currently taking medications that alter CYP3A4 metabolism of glucocorticoids that the participant is unwilling or unable to stop prior to and during the study period e.g. phenytoin, phenobarbital, rifampicin, rifabutin, carbamazepine, primidone, aminogluethimide, itraconazole, ketoconazole, ciclosporin or ritonavir.
* Pregnancy, taking the oral contraceptive pill, or oral oestrogen replacement therapy due to the effects on cortisol binding globulin levels and determination of prednisolone levels. Transdermal oestrogen replacement is permitted. Females of child-bearing age will be asked to provide a urine sample for a pregnancy test at each visit.
* Diagnosis of growth hormone deficiency, untreated
* History of any medical, psychological or other condition, or use of any medications, including over-the-counter products, which, in the opinion of the investigators, would either interfere with the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with either primary or secondary adrenal insufficiency who are currently receiving glucocorticoid replacement therapy with hydrocortisone or prednisolone.
  Healthy volunteers will serve as positive controls.
  Patients on high (anti-inflammatory) doses of steroids for any other medical condition will serve as positive controls.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-04-02 (Estimated); Study Completion 2021-04-02 (Estimated)

PRIMARY OUTCOMES:
Osteocalcin | Single time point for controls. Steroid replacement patients will have been on at least 4 months of stable therapy.
  Assesses bone health of each group by comparing total osteocalcin and undercarboxylated osterocalcin

SECONDARY OUTCOMES:
P1NP | Single time point for controls. Steroid replacement patients will have been on at least 4 months of stable therapy.
  Assesses bone health of each group by comparing P1NP
NTX | Single time point for controls. Steroid replacement patients will have been on at least 4 months of stable therapy.
  Assesses bone health of each group by comparing NTX
Heart Rate | Single time point for controls. Steroid replacement patients will have been on at least 4 months of stable therapy.
  recording observations- heart rate
Blood pressure | Single time point for controls. Steroid replacement patients will have been on at least 4 months of stable therapy.
  recording observations- blood pressure
Waist-Hip circumference | Single time point for controls. Steroid replacement patients will have been on at least 4 months of stable therapy.
  recording observations- Waist-Hip circumference ratios
Lipid profile (Total cholesterol, HDL, LDL and triglycerides) | Single time point for controls. Steroid replacement patients will have been on at least 4 months of stable therapy.
  measuring biochemical indicators of cardiovascular risk: total cholesterol, HDL, LDL and triglycerides
High sensitivity CRP | Single time point for controls. Steroid replacement patients will have been on at least 4 months of stable therapy.
  measuring biochemical indicators of cardiovascular risk: high sensitivity CRP
Glucose | Single time point for controls. Steroid replacement patients will have been on at least 4 months of stable therapy.
  measuring glucose
HbA1c | Single time point for controls. Steroid replacement patients will have been on at least 4 months of stable therapy.
  measuring HbA1c
Infection rates and severity | Single time point for controls. Steroid replacement patients will have been on at least 4 months of stable therapy.
  assessed by completion of the German National Cohort Questionnaire (GNCQ), questionnaires will cover socio-economic and socio-demographic factors, medical history, use of medications and health care, lifestyle factors, and questions related to environmental and occupational factors
Wellbeing | Single time point for controls. Steroid replacement patients will have been on at least 4 months of stable therapy.
  the short form health survey-36 (SF-36)

CONTACTS AND LOCATIONS:
Overall Officials: Karim Meeran, MBBS BSc MD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There are currently no plans to share individual data with other researchers